CLINICAL TRIAL: NCT05936541
Title: Modulation of Bifidocentric Dysbiosis Through Bifidobacterium Bifidum PRL2010 Supplementation in Caesarian-born Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-10/05/2022
Record Dates: First submitted 2023-05-30; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Disbiosis
MeSH Terms: conditions — Dysbiosis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Probiotic Bifidobacterium Bifidum PRL2010
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Bifidobacterium Bifidum PRL2010 (Experimental): Participants in this group will receive probiotic Bifidobacterium Bifidum PRL2010 supplementation from the time of discharge to a daily for the 6 months
  Interventions: Dietary Supplement: Probiotic Bifidobacterium Bifidum PRL2010
- Control (Active Comparator): Participants in this group will not receive probiotic probiotic supplementation
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: Probiotic Bifidobacterium Bifidum PRL2010 — Probiotic supplement
  Arms: Probiotic Bifidobacterium Bifidum PRL2010
Other: Control group — No probiotic supplementation
  Arms: Control

SUMMARY:
This study is aimed to manipulate the composition of the intestinal flora of the infants born by caesarian section through the administration of the probiotic strain "Bifidobacterium bifidum PRL 2010", in order to evaluate its effects on gut dysbiosis during the first 6 month of life.

DETAILED DESCRIPTION:
There has been increasing interest in the field of human microbiome, considering its impact on health and diseases. The gastrointestinal tract represents the most heavily inhabited organ with microorganisms, counting 10 times the total number of human cells; for this reason, the gut microbiome has recently been referred as a proper organ. Intestinal microbial composition is unique for each individual and it is influenced by numerous factors, of which delivery mode is an important one with gestational age of the newborn, type of feeding and intrapartum or neonatal antibiotic therapy. Recent reports suggest that dysbiosis secondary to delivery mode affects the subsequent regulation of immune response and may be associated with several pathologic conditions, for example allergic diseases or obesity. Moreover, gut microbiome seems to impact on neurodevelopment during first six months of life. Bifidobacteria is the most represented group of intestinal microbiota in the newborn, followed by Enterobacteria, and it plays an important role in the infant gut. This includes the fundamental function performed by Bifidobacterium bifidum: it supplies the nutritional material to the rest of the microbial community, particularly Bifidobacterium breve and Bifidobacterium longum infantis that are the other typical bifidobacteria of the newborn. It is a powerful metabolizer of the intestinal mucus and the HMOs (Human Milk Oligosaccharides) present in breast milk. Thanks to its exocitable enzymes, the degradative catabolism occurs in the intestinal environment. Thus, B. bifidum favour the increase in intestinal richness and biodiversity (9), which correlates with the host's state of health. However, bifidobacteria is reduced in infants born by cesarean delivery.

Aim of the study is to assess if the Bifidobacterium Bifidum PRL2010 supplementation effectively ameliorat bifidocentric dysbiosis due to the delivery mode and we want to confirm this by analyzing fecal microbiota in caesarean birth infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants born by caesarian delivery
* Parents informed written consent

Exclusion Criteria

* Suspension of the administration of the probiotic strain for a period of time exceeding 7 days
* Interruption of the administration of the probiotic strain before the completion of the sixth month
* Replacement of Bifidobacterium bifidum PRL2010 with another strain
* Refusal to collect the fecal sample expressed by parents
* Major congenital birth deformities
* Acute illness at enrollment
* Any condition affecting food intake or metabolism
* Maternal mental and psychosomatic diseases

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with disease | up to 6 months
  Number of participants with skin, respiratory and gastrointestinal diseases assessed with a questionnaire submitted to parents

SECONDARY OUTCOMES:
Variation in children gut microbiota composition | up to 6 months
  Variation in gut microbiota composition of children born by caesarean section assessed by faecal colonic microbiota analysis with 16S rRNA technology

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatology and Neonatal Intensive Care Unit of Santa Maria Goretti Hospital, Latina, Italy